CLINICAL TRIAL: NCT06790251
Title: Creation, Management and Analysis of a National Database of Patients With Multiple Endocrine Neoplasia Type 1 (MENNET1 Database)
Brief Title: Institution of an Italian Multicenter Database of Patients With Multiple Endocrine Neoplasia Type 1 (MENNET1 Database)
Status: Not yet recruiting | Type: Observational
Sponsor: F.I.R.M.O. - Fondazione Italiana Ricerca sulle Malattie dell'Osso - Ente del Terzo Settore (Other)
Responsible Party: Sponsor
Other Study IDs: 23922_oss
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Multiple Endocrine Neoplasia Type 1
Keywords: Multiple Endocrine Neoplasia Type 1; Retro-prospective clinical data collection; Database of patients
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with MEN1 syndrome: Male and female patients of any age, who are diagnosed with multiple endocrine neoplasia type 1 (MEN1), including genetic, clinical and/or familiar diagnosis.
  This observational study does not include any type of intervention.

SUMMARY:
The goal of this observational study is to create, manage and analyze a retro-prospective multicenter national database of patients diagnosed with multiple endocrine neoplasia type 1 (MEN1) syndrome (including genetic, clinical and/or familiar diagnosis), aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, and therapeutic data in a relatively high number of patients with this rare inherited endocrine tumor syndrome in Italy.

The study will include 33 specialist clinical centers of endocrinology, pediatric endocrinology, pediatrics, and endocrine surgery, located throughout the Italian territory, and to which patients refer from all the 20 regions of Italy.

Data will be collected over time, both in retrospective and prospective manners, during the 10-year average duration of the study, starting from the recruiting visit (basal visit) and then during each follow-up visits patients will undergo for the control of disease at the recruiting clinical centers, allowing for an epidemiological evaluation of prevalence and incidence of MEN1 in Italy, collecting detailed clinical history of the disease in enrolled patients, and refining and deepening medical knowledge in the field of this rare inherited endocrine tumor syndrome, and, thus, to be able to define optimal tailored diagnostic, clinical, and therapeutic management of patients, improving their quality of life.

Collected data will include both the most classic traits of the pathology and the less common ones.

The main aspects this observational study aims to assess and clarify are:

1. Evaluation of prevalence and incidence of MEN1 in Italy.
2. Clinical characterization of MEN1 phenotypes, through both cross-sectional and longitudinal analyses of collected data, and also based on MEN1 mutation types and location.
3. Evaluation of the over time prevalence of bone mass loss, osteopenia, osteoporosis and fragility fractures in patients with MEN1, with and without primary hyperparathyroidism, globally and also based on gender and age.
4. Over time evaluation of responses to surgical and pharmacological therapies in in patients MEN1.
5. Evaluation of dietary habits in MEN1 patients, by filling out a specific questionnaire at the time of the study recruitment.
6. Evaluation of quality of life and accessibility to specialist medical centers and to surgical and pharmacological therapies on the Italian territory by patients affected by MEN1 syndrome, globally and according to the region of residence, by filling out a specific self-evaluation questionnaire at the time of the study recruitment.

The study will include a single cohort of female and male patients of any age, diagnosed with MEN1 syndrome (including either genetic, clinical and/or familiar diagnosis). The study does not include either any control group/comparison group or healthy volunteers.

The study itself does not involve any medical intervention or drug administration. Surgical and pharmacological treatments for which data on response to therapy will be collected in the database, are those commonly employed for the control/treatment of MEN1 tumors and related symptoms, regardless of patients' inclusion in this observational study.

DETAILED DESCRIPTION:
1. Background and rationale Multiple endocrine neoplasia type 1 (MEN1) is a rare congenital endocrine tumor syndrome characterized by the development of multiple tumors, both benign and malignant, affecting specific neuroendocrine tissues, in particular the parathyroid glands, the anterior pituitary gland, the pancreas, the duodenum, and, more rarely, the adrenal glands, the thymus and the lung/bronchi. The clinical presentation of the disease is extremely variable and includes the combination of over 20 different endocrine and non-endocrine tumors and lesions. The clinical phenotype also differs among members of the same family, and in presence of the same MEN1 gene mutation.

   The incidence is estimated at approximately 1/30,000, with no differences between genders, nor geographic and ethnic prevalence.

   MEN1 syndrome is caused by germline mutations that inactivate the MEN1 tumor suppressor gene (11q13), which encodes the nuclear protein menin, with autosomal dominant inheritance. The mutated copy of the gene is inherited from the affected parent (in over 90% of cases), or, in very rare cases (less than 10%), generated de novo at the embryonic level, and gives the carrier a 100% penetrance to develop the syndrome after the age of 50 years.

   Subjects affected by MEN1 and subjects carrying a MEN1 gene mutation, even if still asymptomatic, must undergo a rigorous program of diagnostic, biochemical and instrumental screening, annually or every two years depending on the tests, throughout their lives, in order to ensure the earliest possible diagnosis of tumors and equally early therapeutic intervention, aimed at reducing morbidity and mortality and improving the quality of life. Accuracy in the differential diagnosis of the syndrome, as well as early diagnosis of tumors, are two fundamental prognostic factors, especially for malignant tumors associated with MEN1, which still cause approximately 30% of deaths.

   The therapy consists of both surgical resection of tumors and specific pharmacological therapies aimed at reducing the growth of functioning and non-functioning tumors or controlling excessive hormone secretion by functioning neuroendocrine tumors.

   Implementing and detailing as much as possible the knowledge on the epidemiology, clinical and therapeutic history, primary and secondary manifestations of MEN1 syndrome, diagnostic techniques, and the response to therapies performed, in a transversal and longitudinal manner, with constant follow-up assessments of patients, also including aspects generally not included in the assessments of this pathology for a long time, such as metabolism and bone health and renal function, is essential not only to improve the clinical management of the individual patient, but also to allow better planning of social, political and health interventions for this pathology and, overall, to improve the quality and life expectancy of patients.

   For this reason, it is extremely important to create a multicenter national database, such as the one proposed by this study, which is able to collect a relatively high number of patients affected by MEN1, whose cases are carefully studied in every aspect, both retrospectively and prospectively, following the course of the disease over time.

   A previous Italian database on MEN1 (MENNET) was established in 2016 and allowed to collect, between 2016 and 2018, over 500 cases of MEN1 patients and/or carriers of mutations on the MEN1 gene from 14 Italian Endocrinological Clinical Centers, located in 9 regions and 11 different cities of the entire peninsula. The analysis of the data collected in the original MENNET database allowed two important publications on clinical and genetic aspects of MEN1. However, this database was exclusively retrospective, with clinical data collection limited exclusively to the time of inclusion in the study and no prospective longitudinal collection of follow-up clinical data was foreseen. The original MENNET database did not include the collection of patients' follow-up clinical data, and only allowed for an epidemiological evaluation and a cross-sectional observational analysis of the data collected at the time of inclusion in the study. To overcome this limitation and to have a longitudinal evaluation of MEN1 syndrome in Italy, this clinical study involves the establishment of a retro-prospective multicenter national database on MEN1 syndrome (MENNET1) that will allow the collection of a case history of patients affected by MEN1 and/or carriers of mutations on the MEN1 gene, whose clinical cases will be studied in detail and also followed over time (follow-up visits), allowing not only to have epidemiological data and perform cross-sectional analyses of the collected data, but also to be able to perform longitudinal analyses of the data, with particular attention to the response to therapies and quality of life.
2. Study population The study will include a single cohort of female and male patients of any age, diagnosed with MEN1 syndrome. The diagnosis of MEN1 syndrome will be considered in subjects with one or more of the following characteristics: 1) presence of at least two of the three main tumors characteristic of MEN1 syndrome (parathyroid adenoma, anterior pituitary adenoma, pancreatic neuroendocrine tumor/duodenal gastrinoma), 2) presence of one of the three main tumors characteristic of MEN1 syndrome and at least one first-degree relative affected by MEN1, 3) presence of a germline mutation on the MEN1 gene.

   The study does not include either any control group/comparison group or healthy volunteers.

   Based on the previous experience with the MENNET database, we can estimate to be able to include in the study at least 600 patients affected by MEN1 during the 10 years of the study.
3. Study design and setting Non-profit, multicenter, national, retro-prospective, observational study, consisting in the design, creation, management and analysis of an Italian database of patients with MEN1.

   The study will have an average duration of 10 years. The enrollment of MEN1 patients, the inclusion in the database with retrospective collection of their clinical data, and the subsequent prospective collection of clinical follow-up data will take place throughout the entire duration of the study. For the retrospective collection, retrospective data on MEN1 syndrome will be retrieved from patient's medical records, at the time of the medical visit that the patient will carry out at the Clinical Center for the evaluation of his/her disease, regardless of inclusion in this study. Prospective data relating to MEN1 follow-up will be collected during the subsequent medical follow-up visits, scheduled for each patient as part of the clinical management of his/her clinical condition, regardless of inclusion in this study.

   Being an observational study, this study itself does not involve the administration of any drug, nor the use of any medical device, nor does it involve additional medical visits, clinical analyses or care procedures in addition to those conventionally scheduled for the clinical and therapeutic management of patient affected by MEN1. No participant biospecimens of any type will be collected and retained to perform this study. Surgical and pharmacological treatments for which data on response to therapy will be collected in the database, are those usually employed in MEN1 patients for the control/treatment of MEN1 tumors and related symptoms, regardless of their inclusion in this observational study.

   All data will be collected anonymously, and they will be analyzed as aggregates. Data collected in the database will be, first, processed using descriptive statistics, such as frequency tables for categorical data, median and quartiles for quantitative data on ordinal scales and mean and standard deviation for quantitative data on metric scales. Secondly, the correlations between variables will be evaluated using the Pearson correlation index in the case of continuous variables and the chi-square test for categorical variables.
4. Data and variables

Data collected in the database will include (if available in patient's medical records and part of the normal clinical and therapeutic management of patient regardless of inclusion in this study):

* Demographics (sex, year of birth)
* Age at diagnosis/onset of MEN1
* Personal clinical history of MEN1
* Family history of MEN1 in first-degree relatives
* Presence of comorbidities
* Result of the genetic testing for MEN1 gene
* Clinical manifestations of the diseases (i.e MEN1-related tumors and other associated, common and rare, clinical manifestations)
* Dual-energy x-ray absorptiometry (DXA) evaluation of bone status (at baseline and follow-up visits)
* History of fragility fractures
* Biochemical measurements of parameters of parathyroid function, bone and mineral metabolism and renal function (at baseline and follow-up visits)
* Surgical interventions (procedure, post-operative outcomes, possible complications, persistence and/or recurrence of disease after surgery)
* Pharmacological therapies (drug, duration, posology)
* Disease-related morbidity and mortality

Moreover, the study will collect, at the time of study recruiting, the following data:

* Patient's dietary habits, collected through the administration of a questionnaire specifically designed for MEN1 patients, which includes data on alcohol and coffee consumption, calcium intake, consumption of antioxidant foods (i.e fruit, dried fruit, vegetables, green tea, foods rich in vitamin C and/or vitamin E, etc), consumption of animal-derived proteins, consumption of refined sugars and high glycemic index foods, consumption of foods rich in oxalates, consumption of processed foods rich in saturated fats
* Self-evaluation of quality of life (i.e self-evaluation of how MEN1 syndrome affects normal daily activities at home, outside and at work, and how it interferes with relationships with other people) and evaluation of accessibility to specialist medical centers and to surgical and pharmacological therapies on the Italian territory. All assessed through a specifically designed questionnaire for MEN1 patients

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MEN1 syndrome (including either genetic, clinical and/or familiar diagnosis)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of female and male patients of any age, diagnosed with MEN1 syndrome. The diagnosis of MEN1 syndrome will be considered in subjects with one or more of the following characteristics: 1) presence of at least two of the three main tumors characteristic of MEN1 syndrome (parathyroid adenoma, anterior pituitary adenoma, pancreatic neuroendocrine tumor/duodenal gastrinoma), 2) presence of one of the three main tumors characteristic of MEN1 syndrome and at least one first-degree relative affected by MEN1, 3) presence of a germline mutation on the MEN1 gene.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence evaluation | Through study completion, an average of 10 years
  Evaluation of prevalence and incidence of MEN1 in Italy
Clinical characterization of MEN1 phenotypes | Through study completion, an average of 10 years
  Clinical characterization of MEN1 phenotypes, through both cross-sectional and longitudinal analyses of collected data, and also based on MEN1 mutation types and location
Bone fragility in patients with MEN1 | Through study completion, an average of 10 years
  Evaluation of the over time prevalence of bone mass loss, osteopenia, osteoporosis and fragility fractures in patients with MEN1, with and without primary hyperparathyroidism, globally and also based on gender and age
Therapy response in MEN1 patients | Through study completion, an average of 10 years
  Over time evaluation of responses to surgical and pharmacological therapies in patients MEN1
Dietary habits in MEN1 patients | Through study completion, an average of 10 years
  Collection of data on dietary habits in MEN1 patients, by filling out a specific questionnaire at the time of the study recruitment, to assess whether patients take in sufficient nutrients that can have a protective effect on the development of tumors (i.e. antioxidants), or beneficial effect on bone health (i.e. calcium and vitamin D), or, on the contrary, they take in excessive quantities of substances that can facilitate the risk of tumors (i.e. animal-derived proteins, refined sugars and high glycemic index foods, processed foods rich in saturated fats ), or the risk of kidney stones (i.e. foods rich in oxalates).
  The questionnaire does not include specific scores on a scale.
Quality of life and accessibility to healthcare and cure for MEN1 patients in Italy | Through study completion, an average of 10 years
  Evaluation of quality of life and accessibility to specialist medical centers and to surgical and pharmacological therapies on the Italian territory by patients affected by MEN1 syndrome, globally and according to the region of residence, by filling out a specific self-evaluation questionnaire at the time of the study recruitment. Quality of life will be specifically assessed through patient's self-evaluation of how MEN1 syndrome affects normal daily activities at home, outside and at work, and how it interferes with relationships with other people, by a series of multiple-choice questions that include, each, a scale of 4 value responses: "not at all", "not much", "enough", "very much", in which "not at all" indicates the best outcome and "very much" the worst one.

CONTACTS AND LOCATIONS:
Locations (33):
- Italy (33):
  - Dipartimento di Scienze Cliniche e Biologiche, Università di Torino, UO di Medicina Interna-Endocrinologia AOU San Luigi Gonzaga, Orbassano, Torino
  - Ambulatorio Tumori Neuro-Endocrini, Unità Operativa Complessa di Oncologia Medica Universitaria, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Bari
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, UO Pediatria, Programma di Malattie Endocrino-Metaboliche, Bologna
  - UOC Endocrinologia e Prevenzione e Cura del Diabete, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Dipartimento di Scienze Mediche e Chirurgiche (DIMEC), Alma Mater Studiorum Università di Bologna, Bologna
  - Endocrinologia e Diabetologia, Azienda Ospedaliero-Universitaria di Cagliari, Presidio Ospedaliero Policlinico di Monserrato, Cagliari
  - SC Endocrinologia, Diabetologia e Metabolismo, ASO Santa Croce e Carle, Cuneo
  - UO Endocrinologia e Malattie del Ricambio, Azienda Ospedaliero Universitaria di Ferrara, Sezione di Endocrinologia, Geriatria e Medicina Interna, Dipartimento di Scienze Mediche, Università degli Studi di Ferrara, Ferrara
  - SOD Malattie del Metabolismo Minerale ed Osseo, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Clinica Endocrinologica, Dipartimento di Medicina Interna e Specialità Mediche (DiMI), IRCCS Ospedale Policlinico San Martino, Università di Genova, Genova
  - UOC di Endocrinologia, AOU Policlinico G. Martino, Dipartimento di Patologia Umana DETEV, Università di Messin, Messina
  - Dipartimento di Malattie Endocrino-Metaboliche, IRCCS Istituto Auxologico Italiano, Milan
  - Divisione di Oncologia Medica Gastrointestinale e Tumori Neuroendocrini, IEO, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - SC Endocrinologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Dipartimento di Medicina Clinica e Chirurgia; Unità di Endocrinologia, Diabetologia e Andrologia; Università degli Studi di Napoli Federico II, Napoli
  - Dipartimento di Pediatria, Azienda Universitaria Ospedaliera della Seconda Università degli Studi di Napoli, Napoli
  - UOC di Endocrinologia e Malattie del Metabolismo, AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - SCDU Endocrinologia Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Unità di Chirurgia Endocrina, Dipartimento di Chirurgia, Oncologia e Gastroenterologia, Università di Padova, Padua
  - UOC Endocrinologia, DIMED, Azienda Ospedaliero-Universitaria di Padova, Padua
  - UOSD Tumori Ereditari, Endocrinologia Oncologica, Dipartimento Oncologia, Unità Tumori Ereditari, Istituto Oncologico Veneto (IOV) di Padova, Padua
  - Unità Operativa Endocrinologia 2, Azienda Ospedaliera Universitaria Pisana, Pisa
  - Dipartimento di Medicina Sperimentale, "Sapienza" Università di Roma, Roma - UOC Endocrinologia, Policlinico Umberto I di Roma, Roma
  - Unità di Endocrinologia e Andrologia, Dipartimento di Medicina Clinica e Molecolare, AOU Sant'Andrea, Centro di eccellenza ENETS, Università Sapienza di Roma, Roma
  - UOC Endocrinologia e Diabetologia, Ospedale Pediatrico Bambin Gesù, Roma
  - UOC di Endocrinologia, Diabetologia e Andrologia Medica, IRCCS Humanitas Research Hospital, Rozzano
  - Donatello Bone Clinic, Casa di Cura Villa Donatello, Sesto Fiorentino
  - Endocrinologia Pediatrica Ospedale Infantile regina Margherita-Dipartimento di Scienze di Sanità Pubblica e Pediatriche, Università degli studi di Torino, Torino
  - SCDU Endocrinologia Diabetologia e Malattie del Metabolismo, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - SCDU Endocrinologia Oncologica, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - SOC Endocrinologia, Azienda Sanitaria-Universitaria Friuli Centrale, Udine
  - Istituto del Pancreas, Azienda Ospedaliera Universitaria Integrata Verona Policlinico G.B Rossi, Verona
  - UOS di Endocrinologia, Policlinico GB Rossi, Azienda Ospedaliera Universitaria Integrata di Verona, Verona

REFERENCES:
- [Background] Marini F, Giusti F, Fossi C, Cioppi F, Cianferotti L, Masi L, Boaretto F, Zovato S, Cetani F, Colao A, Davi MV, Faggiano A, Fanciulli G, Ferolla P, Ferone D, Loli P, Mantero F, Marcocci C, Opocher G, Beck-Peccoz P, Persani L, Scillitani A, Guizzardi F, Spada A, Tomassetti P, Tonelli F, Brandi ML. Correction to: Multiple endocrine neoplasia type 1: analysis of germline MEN1 mutations in the Italian multicenter MEN1 patient database. Endocrine. 2018 Oct;62(1):234-241. doi: 10.1007/s12020-018-1668-3. PMID 30032405
- [Background] Marini F, Giusti F, Fossi C, Cioppi F, Cianferotti L, Masi L, Boaretto F, Zovato S, Cetani F, Colao A, Davi MV, Faggiano A, Fanciulli G, Ferolla P, Ferone D, Loli P, Mantero F, Marcocci C, Opocher G, Beck-Peccoz P, Persani L, Scillitani A, Guizzardi F, Spada A, Tomassetti P, Tonelli F, Brandi ML. Multiple endocrine neoplasia type 1: analysis of germline MEN1 mutations in the Italian multicenter MEN1 patient database. Endocrine. 2018 Oct;62(1):215-233. doi: 10.1007/s12020-018-1566-8. Epub 2018 Mar 1. PMID 29497973
- [Background] Giusti F, Cianferotti L, Boaretto F, Cetani F, Cioppi F, Colao A, Davi MV, Faggiano A, Fanciulli G, Ferolla P, Ferone D, Fossi C, Giudici F, Gronchi G, Loli P, Mantero F, Marcocci C, Marini F, Masi L, Opocher G, Beck-Peccoz P, Persani L, Scillitani A, Sciortino G, Spada A, Tomassetti P, Tonelli F, Brandi ML. Multiple endocrine neoplasia syndrome type 1: institution, management, and data analysis of a nationwide multicenter patient database. Endocrine. 2017 Nov;58(2):349-359. doi: 10.1007/s12020-017-1234-4. Epub 2017 Jan 28. PMID 28132167